CLINICAL TRIAL: NCT05406297
Title: Impact of Trimethylamine N-oxide (TMAO) Serum Levels on Index of Microcirculatory Resistance (IMR) in Patients Diagnosed With ST-Elevation Myocardial Infarction (STEMI)
Brief Title: Impact of TMAO Serum Levels on Hyperemic IMR in STEMI Patients
Acronym: TAMIR
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Università degli Studi di Brescia (Other); Kreiskrankenhaus Rotenburg (Unknown)
Responsible Party: Principal Investigator, Ali Aldujeli, Cardiovascular disease consultant, Lithuanian University of Health Sciences
Other Study IDs: LUHSKC-176
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Microvascular Coronary Artery Disease
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pressure-temperature sensor guidewire-based measurement — In brief, a 6-F angioplasty guiding catheter without side-holes will be used first used to engage the left main coronary artery. A pressure-temperature sensor guidewire ( PressureWire™ X Guidewire) will be used for physiology measurements including IMR measurements.
  Pressure measurement from the wire was first equalized with that of the guiding catheter. Then the pressure sensor will be positioned two-thirds of the way down the LAD artery. Intracoronary nitroglycerin will be administered (100 to 200 μg). Hyperemia will be induced with adenosine intracoronary injections.

SUMMARY:
Trimethylamine N-oxide (TMAO) is a gut microbiota-dependent metabolite of dietary choline, L-carnitine, and phosphatidylcholine-rich foods. On the basis of experimental studies and patients with prevalent disease, elevated plasma TMAO may increase risk of atherosclerotic cardiovascular disease (ASCVD). However, to our knowledge, no data is available on its impact on coronary microcirculation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with STEMI
2. Availability of non- left anterior descending artery (LAD) non culprit lesion, which is planned for a staged Percutaneous coronary intervention (PCI)

Exclusion Criteria:

1. patient undergoing cardiopulmonary resuscitation;
2. patients with a history of old myocardial infarction or history of coronary artery bypass grafting (CABG) or Percutaneous coronary intervention PCI
3. Patients with signs of chronic infection, prolong usage of corticosteroids or compromised immune system
4. patients had thrombolysis before primary Percutaneous coronary intervention (pPCI)
5. had contraindication of adenosine triphosphate (ATP);
6. had a history of liver or renal function dysfunction
7. Patients with dementia
8. Patients being referred to CABG after primary PCI
9. unable to provide informed consent;
10. had pregnancy or life span < 1 year.
11. Presence of sever structural valvular heart disease
12. Presence of significant left main disease
13. Unability to measure the index of microcirculatory resistance due to (death or retraction from the study ...etc)
14. Inability to perform successful PCI

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a prospective, cohort study, conducted in the Hospital of the Lithuanian University of Health Sciences Kaunas Clinics.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Index of microcirculatory resistance | 3 months
  The index of microcirculatory resistance (IMR) will be detected using PressureWire™ X Guidewire

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 3 months
  left ventricular ejection fraction will be assessed via echocardiography imaging using Simpson's biplane method.
major adverse cardiovascular events (MACE) | up to 1 year
  . MACE was defined as follows: cardiovascular death, non-fatal myocardial infarction, target vessel revascularization, recurrent hospitalization due to decompensated heart failure, and stroke (ischemic or hemorrhagic).

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Aldujeli, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aldujeli A, Tsai TY, Haq A, Tatarunas V, Garg S, Hughes D, Ciapiene I, Unikas R, Sharif F, Lesauskaite V, Onuma Y, Serruys PW. The association between trimethylamine N-oxide levels and coronary microvascular dysfunction and prognosis in patients with ST-elevation myocardial infarction. Atherosclerosis. 2024 Nov;398:118597. doi: 10.1016/j.atherosclerosis.2024.118597. Epub 2024 Sep 12. PMID 39316928
- [Derived] Tsai TY, Aldujeli A, Haq A, Knokneris A, Briedis K, Hughes D, Unikas R, Renkens M, Revaiah PC, Tobe A, Miyashita K, Sharif F, Garg S, Onuma Y, Serruys PW. The Impact of Microvascular Resistance Reserve on the Outcome of Patients With STEMI. JACC Cardiovasc Interv. 2024 May 27;17(10):1214-1227. doi: 10.1016/j.jcin.2024.03.024. Epub 2024 May 14. PMID 38752970
- [Derived] Aldujeli A, Tsai TY, Haq A, Tatarunas V, Knokneris A, Briedis K, Unikas R, Onuma Y, Brilakis ES, Serruys PW. Impact of Coronary Microvascular Dysfunction on Functional Left Ventricular Remodeling and Diastolic Dysfunction. J Am Heart Assoc. 2024 May 7;13(9):e033596. doi: 10.1161/JAHA.123.033596. Epub 2024 Apr 30. PMID 38686863
- [Derived] Aldujeli A, Haq A, Tsai TY, Grabauskyte I, Tatarunas V, Briedis K, Rana S, Unikas R, Hamadeh A, Serruys PW, Brilakis ES. The impact of primary percutaneous coronary intervention strategies during ST-elevation myocardial infarction on the prevalence of coronary microvascular dysfunction. Sci Rep. 2023 Nov 16;13(1):20094. doi: 10.1038/s41598-023-47343-x. PMID 37973856